CLINICAL TRIAL: NCT03427684
Title: Phase I Study of Hypo-fractionated Neoadjuvant Radiotherapy for Locally Advanced Gastric Cancer
Brief Title: Study of Hypo-fractionated Neoadjuvant Radiotherapy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LI Ning, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMS-GIRO-G005
Record Dates: First submitted 2018-01-28; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer; Chemoradiation
Keywords: Gastric cancer; Chemo-radiotherapy; Phase I study; Hypo-fractionated radiotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo-fractionated radiotherapy (Experimental): Hypo-fractionated neoadjuvant radiotherapy concurrent with S1 chemotherapy for local advanced gastric cancer
  Interventions: Radiation: Hypo-fractionated radiotherapy; Drug: S1

INTERVENTIONS:
Radiation: Hypo-fractionated radiotherapy — Hypo-fractionated radiotherapy with fraction >2Gy .
Drug: S1 — S-1 80mg/m2/day, orally intake on radiotherapy days.

SUMMARY:
Gastric cancer is one of the most common malignant tumors in China, and the incidence and mortality rate are second in malignant tumors. The treatment of gastric cancer need integrated multidisciplinary treatment, and surgery is the only possible curative method for gastric cancer at present. Previous studies have reported that neoadjuvant chemoradiotherapy can downstage primary tumor to increase radical resection rate in order to improve the long-term prognosis of advanced gastric cancer. However, there is no study on the application of hypo-radiotherapy to neoadjuvant radiotherapy in gastric cancer. The aim of this study was to observe the maximum tolerated dose (MTD) and dose limited toxicity (DLT) of hypo-fractionated radiotherapy for locally advanced gastric cancer.

DETAILED DESCRIPTION:
After enrolled in this study, the patient was first treated with radiotherapy, concurrent with oral S-1 80mg/m2/day, on radiotherapy days. 3 weeks after the end of radiotherapy, patients treated with neoadjuvant chemotherapy with oxaliplatin and S-1. Oxaliplatin is given on dose of 130mg/m2 iv on day 1; S-1 on 40-60mg po BID on day 1-14, oral. Imaging evaluation was performed 3 weeks after neoadjuvant treatment. The radical operation and surgical procedure were determined on MDT discussion. Non-operable patients continue with 3 cycles of chemotherapy, and the chemotherapy regimen can be changed. A 3 cycle of SOX adjuvant chemotherapy was performed after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T3-4N+M0
* Gastric cancer or Siewert II/III esophagogastric junction carcinoma;
* Pathologically confirmed adenocarcinoma;
* 18-75 years old, male or female;
* Karnofsky score >= 70;
* White blood cell count >= 4 x 109 / L; platelet count >= 100 x109/L; serum creatinine =< 1 x upper limit of normal, total bilirubin =< 1 x upper limit of normal, alanine aminotransferase and aspartate aminotransferase =< 2.5 x upper limit of normal, alkaline phosphatase =< 5 x upper limit of normal.

Exclusion Criteria:

* Any chemotherapy or radiotherapy history before enrollment
* Siewert I EGJ cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose AND Dose limited toxicity | From date of enrollment until one month after chemo-radiotherapy
  To assess maximum tolerated dose and dose limited toxicity of hypo-fractionated neoadjuvant radiotherapy

SECONDARY OUTCOMES:
Response rate | From date of enrollment until surgery, assessed up to 2 months
  To evaluate the pathological response rate of gastric cancer after hypo-fractionated neoadjuvant radiotherapy
2-year disease-free survival | From date of enrollment until the date of first documented progression or date of relapse, whichever came first, assessed up to 24 months
  To evaluate the 2-year disease-free survival of gastric cancer after hypo-fractionated neoadjuvant radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Li N, Xiang X, Zhao D, Wang X, Tang Y, Chi Y, Yang L, Jiang L, Jiang J, Shi J, Liu W, Fang H, Tang Y, Chen B, Lu N, Jing H, Qi S, Wang S, Liu Y, Song Y, Li Y, Zhang L, Jin J. Preoperative versus postoperative chemo-radiotherapy for locally advanced gastric cancer: a multicenter propensity score-matched analysis. BMC Cancer. 2022 Feb 26;22(1):212. doi: 10.1186/s12885-022-09297-7. PMID 35219300
- [Derived] Li N, Wang X, Tang Y, Zhao D, Chi Y, Yang L, Jiang L, Jiang J, Liu W, Tang Y, Fang H, Liu Y, Song Y, Wang S, Jin J, Li Y. A prospective phase I study of hypo-fractionated neoadjuvant radiotherapy for locally advanced gastric cancer. BMC Cancer. 2018 Aug 8;18(1):803. doi: 10.1186/s12885-018-4707-9. PMID 30089457